CLINICAL TRIAL: NCT04671342
Title: Diagnostic Validation of the DreamKit Device Against Polysomnography
Brief Title: DreamKit Diagnostic Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRC_SLE_Sparkle_PSG_2020_10908
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Validation Arm (Experimental): Participants will wear the DreamKit device (test device) while instrumented with polysomnography sensors (gold standard).
  Interventions: Device: DreamKit

INTERVENTIONS:
Device: DreamKit — The DreamKit device is a single-use device intended to aid the diagnosis of sleep-disordered breathing.

SUMMARY:
This study has been developed in order to demonstrate diagnostic efficacy of the DreamKit device against polysomnography.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the diagnostic performance of the DreamKit device against the gold-standard comparator, polysomnography (PSG). Data collection will be completed within a single visit, in which participants will undergo simultaneous measurement using the DreamKit device and in-laboratory PSG.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Fluent in English;
* Able to provide informed consent.

Exclusion Criteria:

* Self-reported habitual sleep duration of <4 hours/night on average ("How many hours sleep do you usually get per night?");
* Circadian phase disorder, shift work, or any other issue/condition that would, in the opinion of the site investigator, reduce the likelihood of obtaining at least four hours of sleep during the overnight study;
* History of allergic reactions to medical adhesives;
* Skin rash or other dermatological condition that would impact correct placement of the DreamKit device and/or PSG sensors, and/or would be exacerbated by the presence of the device or sensors;
* Presence of a pacemaker;
* Severe medical condition (controlled or uncontrolled) that would impede data collection in the opinion of the site investigator, including the requirement for oxygen therapy;
* [for those currently using overnight therapy]: Unwilling to withdraw from overnight therapy for a single night and/or clinically unsuitable to withdraw from overnight therapy in the opinion of the site investigator, with overnight therapy including but not limited to any form of PAP or ventilation, oral device including mandibular advancement devices or mouthguard for bruxism, nasal dilator strips, and/or positional device;
* [for those currently using overnight therapy]: Considered by the site investigator to be at risk of an AE resulting from hypersomnolence the day after the overnight visit, such as a high-risk occupation including but not limited to a pilot or commercial driver;
* An employee, or family member of an employee, of a company that designs, sells, or manufactures sleep related products (including Philips).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Hardy, Study Director — Philips Sleep & Respiratory Care
Locations (7):
- United States (7):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Florida Lung and Sleep Associates, Lehigh Acres, Florida
  - Pulmonary and Critical Care Association of Baltimore, Towson, Maryland
  - Clayton Sleep Institute, Maplewood, Missouri
  - Berks Schuylkill Respiratory Specialists, Wyomissing, Pennsylvania
  - Bogan Sleep Consultants, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total participants that were consented.
Groups:
- DreamKit Device Intervention: Participants will wear the DreamKit device (test device) while instrumented with polysomnography sensors (gold standard).
  DreamKit: The DreamKit device is a single-use device intended to aid the diagnosis of sleep-disordered breathing.
Period: Consented and Screened (Visit 1)
Arm/Group | DreamKit Device Intervention
Started | 306
Completed | 259
Not Completed | 47
Not completed — Screen Failure | 3
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawn by sponsor due to recruitment consideration (CSA patients) | 39
Period: Completed Visit 2 With Evaluable Data
Arm/Group | DreamKit Device Intervention
Started | 259
Completed | 200
Not Completed | 59
Not completed — Unusable device data | 58
Not completed — Unusable PSG data | 1

BASELINE CHARACTERISTICS:
Population: All participants that were consented
Arm/Group | Validation Arm
Number analyzed (Participants) | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data (Sex) available for 297 of 306 participants.
  Participants
    number analyzed (Participants) | 297
    Female | 123
    Male | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data (Ethnicity) available for 297 of 306 participants.
  Participants
    number analyzed (Participants) | 297
    Hispanic or Latino | 45
    Not Hispanic or Latino | 251
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data (Race) available for 300 of 306 participants.
  Participants
    number analyzed (Participants) | 300
    American Indian or Alaska Native | 3
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 29
    White | 262
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Population: Demographic information only available and analyzed for 297 out of 306 participants. All enrollment occurred in the United States.
  participants
    United States: number analyzed (Participants) | 297
    United States | 297

OUTCOME MEASURES:

1. Primary Outcome: Intraclass Correlation Coefficient (ICC) of the Apnea Hypopnea Index
Description: The primary endpoint is the intraclass correlation coefficient (ICC) for absolute agreement between the polysomnography (PSG) apnea-hypopnea index (AHI) and the DreamKit-AHI. The higher ICC indicates higher correlation/agreement between the PSG AHI and DreamKit AHI. The possible range of ICC values is 0 to 1.0. Number was the best option for the measure type because it was a correlation coefficient.
Time Frame: Visit 2 (within six weeks of enrollment)
Population: Completed Visit 2 with evaluable data
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Arm/Group | Validation Arm
Number analyzed (Participants) | 200
intraclass correlation coefficient (ICC) | 0.964 [0.953 to 0.973]

2. Secondary Outcome: Intraclass Correlation Coefficient (ICC) of the Central Apnea Index
Description: The secondary endpoint is the ICC for absolute agreement between the PSG-central apnea index (CAI) and the DreamKit-CAI. The higher ICC indicates higher correlation/agreement between the PSG CAII and DreamKit CAI. The possible range of ICC values is 0 to 1.0. Number was the best option for the measure type because it was a correlation coefficient.
Time Frame: Visit 2 (within six weeks of enrollment)
Population: Completed Visit 2 with evaluable data
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Arm/Group | Validation Arm
Number analyzed (Participants) | 200
intraclass correlation coefficient (ICC) | 0.731 [0.659 to 0.790]

ADVERSE EVENTS:
Time Frame: Throughout the individual's participation in the study, (Visit 1 and Visit 2) and up to 7 days after completing visit 2
Arm/Group | Validation Arm
All-Cause Mortality (participants affected / at risk) | 0/306
Serious Adverse Events (participants affected / at risk) | 0/306
Other Adverse Events (participants affected / at risk) | 7/306
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Validation Arm (N=306)
Side Effects from COVID vaccine (General disorders) | 1 (2)
Upper Airway Dryness alleged from not using their CPAP therapy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mouth/Tongue Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Struck head during PSG (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain due to exercise (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Ear Pain due to Electrode placement (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04671342/Prot_SAP_000.pdf